CLINICAL TRIAL: NCT05275842
Title: Development and Feasibility Testing of an Integrated PTSD and Adherence Intervention Cognitive Processing Therapy-Lifesteps (CPT-L) to Improve HIV Outcomes
Brief Title: CPT-L to Improve Outcomes for Individuals With HIV and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cristina Lopez, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00106801; 1R34MH125706-01A1 (NIH)
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: PTSD; Hiv
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] (Experimental)
  Interventions: Behavioral: Cognitive Processing Therapy- Lifesteps (CPT-L); Behavioral: Lifesteps
- Lifesteps [Group B] (Active Comparator)
  Interventions: Behavioral: Lifesteps

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy- Lifesteps (CPT-L) — CPT-L is designed to help people with HIV and PTSD take their medications as prescribed. Cognitive Processing Therapy (CPT) uses education and cognitive training to help individuals identify thoughts and feelings about their trauma and gives them tools to help them change unhelpful beliefs. Lifesteps (L) includes education on the need for people with HIV to take their medications as prescribed and what could happen if you do not, as well as gives you tools to help motivate and remind you to take your medications on time.
  Participants will receive a 12-session Cognitive Processing Therapy-Lifesteps (CPT-L) treatment program at the Ryan White clinic. The CPT-L program will be delivered twice a week for 6 weeks. Each session last about 90-minutes.
  Arms: Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A]
Behavioral: Lifesteps — Lifesteps (L) includes education on the need for people with HIV to take their medications as prescribed and what could happen if you do not, as well as gives you tools to help motivate and remind you to take your medications on time.
  Participants will complete one Lifesteps education session. This session lasts about 60 minutes. Participants may attend this session either in-person or over the internet if they have an internet ready device with audio.

SUMMARY:
This study plans to adapt and examine the acceptability and feasibility of an evidence-based PTSD treatment that has reduced other HIV transmission behavior (e.g., sexual risk), Cognitive Processing Therapy (CPT), at an HIV clinic as a strategy to improve HIV outcomes in this population.

DETAILED DESCRIPTION:
The prevalence of trauma exposure, and post-traumatic stress disorder (PTSD) in particular, among individuals living with HIV (30-74%) is higher than the general population (7-10%). Individuals with co-occurring PTSD and HIV are at high-risk for negative HIV-related outcomes, including low adherence to antiretroviral therapy (ART), faster disease progression, more hospitalizations, and almost twice the rate of death, as well as increased mental health problems. In addition to PTSD resulting from traumatic events, such as sexual and physical assault/abuse, negative reinforcement conceptual models suggest that the avoidant behavior (a hallmark symptom of PTSD) tied to HIV status-related PTSD can also contribute to poor ART adherence and to less success of viral suppression (e.g., by avoiding cues, such as ART medications, that serve as reminders of the HIV status). Despite the high rates of persons living with HIV/AIDS (PLWH) who report PTSD - and the poorer HIV patient outcomes among this population versus those without co-occurring PTSD- evaluation of the impact of evidence-based treatment for PTSD among populations living with HIV on HIV outcomes has been highly neglected in clinical research. In other words, no research to date has examined the critical question of whether HIV outcomes can be improved among the large number of PLWH with co-morbid PTSD and related consequences (e.g., substance misuse) by treating PTSD symptoms.

To address this tremendous void in the field, we propose to adapt and examine the acceptability and feasibility of an evidence-based PTSD treatment that has reduced other HIV transmission behavior (e.g., sexual risk), Cognitive Processing Therapy (CPT), at an HIV clinic as a strategy to improve HIV outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals that are 18 years and older
2. Linked with and/or eligible for treatment at a Ryan White clinic in South Carolina.
3. Participant meets clinically significant threshold of DSM-V PTSD criteria as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview.
4. No changes in psychotropic medication within 4 weeks of study enrollment.
5. Able to speak, read, and write English.
6. Meet at least one of the following HIV care criteria:

   1. Diagnosed with HIV in the last 3 months;
   2. Detectable viral load in the last 12 months;
   3. Failed to show up for or missed 1 or more HIV care appointments in the past 12 months;
   4. Last HIV care visit was more than 6 months ago;
   5. Self-reporting less than 90% ART adherence in the past 4 weeks.
7. A score of at least 10 on the Montreal Cognitive Assessment test (MoCA)

Exclusion Criteria:

1. Evidence of significant cognitive impairment as assessed by the Montreal Cognitive Assessment Test (MoCA; in the severe range).
2. Evidence of developmental delays, or pervasive developmental disorder, or active suicidal or homicidal ideations.
3. Evidence of psychotic symptoms (e.g., active hallucinations, delusions, impaired thought processes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lopez, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez C, Baker N, Amaya S, Bisca E, Wilson T, Eckard AR, Moreland A, Resick PA, Safren SA, Danielson CK. Integrated PTSD and Adherence Treatment for People with HIV: Main Findings of a Feasibility Pilot for Cognitive Processing Therapy-Lifesteps (CPT-L). Res Sq [Preprint]. 2025 May 27:rs.3.rs-6567722. doi: 10.21203/rs.3.rs-6567722/v1. PMID 40502775
- [Derived] Lopez CM, Moreland AD, Amaya S, Bisca E, Mujica C, Wilson T, Baker N, Richey L, Eckard AR, Resick PA, Safren SA, Danielson CK. Assessment, Decision, Adaptation, Production, Topical Experts-Integration, Training, and Testing (ADAPT-ITT) Framework to Tailor Evidence-Based Posttraumatic Stress Disorder Treatment for People With HIV to Enhance Engagement and Adherence: Qualitative Results from a Feasibility Randomized Controlled Trial. JMIR Form Res. 2025 Jan 16;9:e64258. doi: 10.2196/64258. PMID 39819749

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A]: Cognitive Processing Therapy- Lifesteps (CPT-L): CPT-L is designed to help people with HIV and PTSD take their medications as prescribed. Cognitive Processing Therapy (CPT) uses education and cognitive training to help individuals identify thoughts and feelings about their trauma and gives them tools to help them change unhelpful beliefs. Lifesteps (L) includes education on the need for people with HIV to take their medications as prescribed and what could happen if you do not, as well as gives you tools to help motivate and remind you to take your medications on time.
  Participants will receive a 12-session Cognitive Processing Therapy-Lifesteps (CPT-L) treatment program at the Ryan White clinic. The CPT-L program will be delivered twice a week for 6 weeks. Each session last about 90-minutes.
  Lifesteps: Lifesteps (L) includes education on the need for people with HIV to take their medications as prescribed and what could happen if you do not, as well as gives you tools to help motivate and remind you to take your medications on time.
  Participants will complete one Lifesteps education session. This session lasts about 60 minutes. Participants may attend this session either in-person or over the internet if they have an internet ready device with audio.
Period: Overall Study
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Started | 20 | 21
Completed | 12 | 17
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Population is denoted as all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B] | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.8) | 40.8 (11.6) | 44.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 14 | 25
  White | 8 | 4 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to:
  Make current (past month) diagnosis of PTSD Make lifetime diagnosis of PTSD Assess PTSD symptoms over the past week.
  Higher scores indicate greater PTSD symptoms.
  units on a scale | 33.5 (8.8) | 37.0 (9.7) | 35.3 (9.3)
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including:
  Monitoring symptom change during and after treatment Screening individuals for PTSD Making a provisional PTSD diagnosis
  Higher scores indicate greater PTSD symptoms.
  units on a scale | 36.8 (12.3) | 42.6 (11.3) | 39.7 (12)
Detectible Viral Load [Count of Participants; unit: Participants] — Population: One participant did not have Viral Load data available in medical record at study baseline.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 9 | 7 | 16
Medication Compliance [Mean (Standard Deviation); unit: Percentage of Doses Taken] — Self reported percentage of medication doses take in the past 30 days. Measured at study baseline. Range 0.0% to 100.0%. Population: Data as collected as a part of the baseline survey and some data is item missing.
  Percentage of Doses Taken
    number analyzed (Participants) | 17 | 17 | 34
    (all) | 90.9 (21.9) | 93.8 (11.5) | 92.4 (17.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Participants
Description: The percentage of participants that were classified as eligible out of all participants that were screened for the purpose of the study.
Time Frame: Study Screening Visit
Population: Screened population
Measure: Count of Participants; unit: Participants
Groups:
- Cohort: flow of participant prior to randomization, noted as the number eligible out of the screened population
Arm/Group | Cohort
Number analyzed (Participants) | 534
Participants | 85

2. Primary Outcome: Percent of Completed Participants
Description: The percentage of participants that were enrolled and completed the study protocol.
Time Frame: 6-week end of study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Number analyzed (Participants) | 20 | 21
Participants | 12 | 17

3. Primary Outcome: Average Number of Enrolled Participants Per Month
Description: The average number of recruited participants per month (across the entirety of the enrollment window).
Time Frame: Approximately 24 months of active recruitment
Population: flow rate of randomized participants during study recruitment
Measure: Mean (Full Range); unit: Participants per month
Arm/Group | Cohort
Number analyzed (Participants) | 41
Participants per month | 1.71 [0 to 6]

4. Secondary Outcome: Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: PTSD symptoms are measured by the CAPS-5 scale, an empirically supported clinician-report instrument. CAPS-5 includes 20 items with a likert scale of 0 (not at all) to 4 (extremely). Scores range from total symptom count of 0-80. Higher scores indicate more severe PTSD symptoms.
Time Frame: These measures will be collected at baseline and the 6 week end of study treatment visit.
Population: analysis population is those who were randomized to study treatment and have data available at the end of study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Number analyzed (Participants) | 11 | 17
units on a scale | 18.5 (15.1) | 29.4 (14.3)

5. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: PTSD symptoms are measured by the PCL-5 scale, an empirically supported self-report instrument. PCL-5 includes 20 items with a likert scale of 0 (not at all) to 4 (extremely). Scores range from total symptom count of 0-80. Higher scores indicate more severe PTSD symptoms.
Time Frame: These measures will be collected at baseline and the 6 week end of study treatment visit.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Number analyzed (Participants) | 11 | 17
units on a scale | 18.5 (20.5) | 33.7 (16.8)

6. Secondary Outcome: Number of Patients With Suppressed Viral Load
Description: Results from standard clinical assays (collected for clinical purposes). An HIV viral load less than 200 will be considered consistent with virologic suppression. The results of a viral load are described as the number of copies of HIV RNA in a milliliter of blood. A viral load of 10,000 would be considered low; 100,000 or above would be considered high.
Time Frame: These measures will be collected at 6 months after enrollment.
Population: those with available viral load data taken between end of study treatment and follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Number analyzed (Participants) | 15 | 13
Participants | 14 | 10

7. Secondary Outcome: Medication Pill Count / Compliance
Description: Self Reported percentage of doses taken during the past 30 days. Range 0.0 - 100.0.
Time Frame: Measure taken at study baseline and at the close of study treatment (6 week visit)
Population: Available data at the close of study treatment (6-week visit)
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
Number analyzed (Participants) | 7 | 13
percentage of doses taken | 99.1 (1.5) | 89.2 (27.1)

ADVERSE EVENTS:
Time Frame: Adverse events are monitored from study enrollment through the completion of 3-month study follow up visit, an average of 3 months.
Arm/Group | Cognitive Processing Therapy-Lifesteps (CPT-L) [Group A] | Lifesteps [Group B]
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
Viral load often not collected clinically within time frame of data collection in electronic medical record; method used to collect objective pill count produced 66% missing so it could not be analyzed or summarized; recruitment challenges with staff turnover, institutional barriers to specifying information on project flyers, resulting in many eligibility screens that did not meet criteria; recruitment barriers getting into certain clinics who had not collaborated on research projects before.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT05275842/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT05275842/ICF_002.pdf